CLINICAL TRIAL: NCT02392039
Title: Randomized, Placebo Controlled Study of Loratadine for Pegfilgrastim Induced Bone Pain in Patients With Aggressive Lymphoma
Brief Title: Study of Loratadine for Pegfilgrastim Induced Bone Pain in Patients With Aggressive Lymphoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-0880; NCI-2015-00592 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Lymphoma
Keywords: Lymphoma; Diffuse Large B-cell Lymphoma; Mantle Cell Lymphoma; Grade 3B Follicular Lymphoma; Burkitt Lymphoma; Peripheral T cell Lymphoma NOS; NK/T cell Lymphoma; Transformed Lymphoma; Aggressive lymphoma; Bone pain; Pegfilgrastim; Neulasta; PEG-G-CSF; Loratadine; Placebo; Sugar pill; Questionnaires; Surveys
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma, T-Cell; Lymphoma, Extranodal NK-T-Cell | interventions — pegfilgrastim; pegylated granulocyte colony-stimulating factor, human; Loratadine; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - Loratadine (Experimental): Pegfilgrastim 6 mg subcutaneously between 24 and 72 hours after completion of chemotherapy once per 21 day cycle.
  Cycle 1 and 3:
  Loratadine 10 mg by mouth daily, starting on the day of Pegfilgrastim administration and continuing for a total of 7 days.
  Cycle 2 and 4:
  Placebo by mouth daily, starting on the day of Pegfilgrastim administration and continuing for a total of 7 days.
  Three questionnaires completed about bone pain and quality of life. These are completed before Pegfilgrastim received during Cycles 1 - 4 (and if participant has pain, during Cycles 6 - 7), on Day 7, and 8 weeks after last dose of study drugs.
  Interventions: Drug: Pegfilgrastim; Drug: Loratadine; Other: Placebo; Behavioral: Questionnaires
- Group 2 - Placebo (Experimental): Pegfilgrastim 6 mg subcutaneously between 24 and 72 hours after completion of chemotherapy once per 21 day cycle.
  Cycle 1 and 3:
  Placebo by mouth daily, starting on the day of Pegfilgrastim administration and continuing for a total of 7 days.
  Cycle 2 and 4:
  Loratadine 10 mg by mouth daily, starting on the day of Pegfilgrastim administration and continuing for a total of 7 days.
  Three questionnaires completed about bone pain and quality of life. These are completed before Pegfilgrastim received during Cycles 1 - 4 (and if participant has pain, during Cycles 6 - 7), on Day 7, and 8 weeks after last dose of study drugs.
  Interventions: Drug: Pegfilgrastim; Drug: Loratadine; Other: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Pegfilgrastim — 6 mg subcutaneously between 24 and 72 hours after completion of chemotherapy once per 21 day cycle.
  Other Names: Neulasta; PEG-G-CSF
Drug: Loratadine — Group 1 - Cycles 1 and 3: Loratadine 10 mg by mouth daily, starting on the day of Pegfilgrastim administration and continuing for a total of 7 days.
  Group 2 - Cycle 2 and 4: Loratadine 10 mg by mouth daily, starting on the day of Pegfilgrastim administration and continuing for a total of 7 days.
Other: Placebo — Group 1 - Cycle 2 and 4: Placebo by mouth daily, starting on the day of Pegfilgrastim administration and continuing for a total of 7 days.
  Group 2 - Cycle 1 and 3 : Placebo by mouth daily, starting on the day of Pegfilgrastim administration and continuing for a total of 7 days.
  Other Names: Sugar Pill
Behavioral: Questionnaires — Three questionnaires completed about bone pain and quality of life. These are completed before Pegfilgrastim received during Cycles 1 - 4 (and if participant has pain, during Cycles 6 - 7), on Day 7, and 8 weeks after last dose of study drugs.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if loratadine can control bone pain caused by pegfilgrastim (a drug given after chemotherapy to help raise white blood cell counts).

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being in either group.

* If you are in Group 1, during Cycles 1 and 3 you will receive loratadine. During Cycles 2 and 4, you will receive a placebo.
* If you are in Group 2, during Cycles 1 and 3 you will receive a placebo. During Cycles 2 and 4, you will receive a loratadine.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

Both groups will receive pegfilgrastim after standard of care chemotherapy.

Neither you nor the study staff will know when you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

Each study cycle is 21 days.

On Day 1 of Cycles 1-6, you will receive pegfilgrastim through a needle under the skin.

On Days 1-7 of Cycles 1-4, you will take loratadine/placebo by mouth 1 time every day.

If you have any bone pain during Cycles 1-4, you will take loratadine on Days 1-7 of Cycles 5 and 6. If you do not have bone pain, you will be off study after Cycle 4.

The study doctor will decide if you need any extra pain medication.

You will be given a diary to write down when you take loratadine/placebo, and to write down the amount and time of any pain medications they need, and to describe the location, severity, and description of the pain you experience.

Study Visits:

During Cycles 1-4 (and if you have pain, during Cycles 6-7), before you receive pegfilgrastim and on Day 7, you will complete 3 questionnaires about your bone pain and how you are feeling. The should take about 20 minutes to complete. If you are not coming into the clinic, you will be asked to mail in the questionnaires and your diary.

Before each cycle starts, blood (about 2-4 teaspoons) will be drawn for routine tests and to test your liver, bone, and kidneys.

On Day 1 of Cycles 2-6, you will have a physical exam, and blood (about 3-4 teaspoons) will be drawn for routine tests.

On Days 7 and 14 of each cycle (+/- 3 days), blood (about 2-4 teaspoons) will be drawn for routine tests.

Length of Study:

You may continue taking the study drugs for up to 18 weeks (6 cycles). You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation in this study will be over after the end-of-study visit.

End-of-Study Visit:

Within 8 weeks after your last dose of study drugs:

* You will have a physical exam.
* You will complete the 3 questionnaires about your bone pain and how you are feeling.
* Blood (about 2-4 teaspoons) will be drawn for routine tests and to test your liver, bone, and kidneys.

This is an investigational study. Loratadine is FDA approved and commercially available for the treatment of seasonal allergies. Pegfilgrastim is FDA approved and commercially available for improvement of chemotherapy-related neutropenia. The use of loratadine to control bone pain is investigational.

Up to 56 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have newly diagnosed, previously untreated Diffuse Large B-cell Lymphoma, Mantle Cell Lymphoma, Grade 3B Follicular lymphoma, Burkitt Lymphoma, Peripheral T cell Lymphoma NOS, NK/T cell Lymphoma, or Transformed lymphoma.
2. Planned to receive chemotherapy for 6 cycles which the treating physician plans to utilize for pegfilgrastim to minimize risk for neutropenic fever, including but not limited to R-CHOP, R-EPOCH, and R-HyperCVAD, CHOP, and SMILE.
3. Age >= 18 years old.
4. ECOG performance status 0-3.
5. Ability to provide informed consent for participation.

Exclusion Criteria:

1. Existing chronic bone pain prior to pegfilgrastim usage.
2. Creatinine clearance of <50ml/minute by Cockcroft Gault equation.
3. Allergy to filgrastim, pegfilgrastim, or Loratadine.
4. Chronic daily usage of antihistamine without an acceptable alternative non-antihistamine medication.
5. Inability to swallow medications.
6. Inability to complete the survey instrumentation accurately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Bone Pain Related Quality of Life (QOL) Measured by FACT-Bone Pain (FACT-BP) Questionnaire | 26 weeks
  FACT-BP (range: 0 - 60) questionnaire used to measure patients bone pain. Participant considered having bone pain if the answer for question BP1 in the FACT-BP questionnaire is >0.

CONTACTS AND LOCATIONS:
Overall Officials: Jason R. Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org